CLINICAL TRIAL: NCT01574300
Title: Collaborative Advanced Stage Tissue Lung Cancer (CASTLE) Network
Acronym: CASTLE
Status: Terminated | Type: Observational
Why Stopped: interim assessment by sponsor
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: VICC THO 09110; CASTLE Study (Other: Adarrio Lung Cancer Institute (ALCMI))
Record Dates: First submitted 2012-03-28; First posted 2012-04-10 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Small Cell Lung Carcinoma
Keywords: Small Cell Lung Cancer (SCLC); Non-Small Cell Lung Cancer (NSCLC); M1A or B NSCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Coal Tar

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biospecimens and biofluids: This is a multi-cohort parallel study in which tumor, plasma and serum samples will be collected prior to the start of any therapeutic intervention for stage IV lung cancer. These biospecimens will be correlated with treatment and clinical data and distributed for peer reviewed research purposes to academic and community centers in the U.S. and Europe.
  The biospecimens collected in CASTLE will be analyzed for a panel of biomarkers, currently including:
  * tumor: epidermal growth factor receptor (EGFR), KRAS (Kirsten RAt Sarcoma) gene and EML4-ALK (echinoderm microtubule-associated protein-like 4 - anaplastic lymphoma kinase) translocations, and EGFR, TS (thymidylate synthase), ERCC1 (excision repair cross-complementing 1) and RRM1 (Ribonucleotide Reductase, M1 Subunit) gene expressions
  * serum: proteomics predictive for EGFR-TKI (tyrosine kinase inhibotors)response
  Interventions: Other: therapeutic interventions

INTERVENTIONS:
Other: therapeutic interventions — All therapeutic interventions are allowed, and their details recorded and correlated with data from the collected biospecimens. Examples would include single or multiple agent chemotherapy or targeted therapeutics

SUMMARY:
The purpose of this study is to facilitate application of the known biomarkers to patients presenting today, and to establish a collection of biospecimens that will be useful for discovering and validating new biomarkers for future use.

DETAILED DESCRIPTION:
Because of the historically poor outcomes of lung cancer patients, suboptimal therapeutic efficacy, and significant side effects of chemotherapy, and the need to choose more efficacious treatment regimens, and patients most likely to benefit from them, there is a need to predict a priori whether an individual patient's tumor will respond to a particular therapeutic agent. However, virtually all lung cancer tumor samples available today are from resection specimens so direct, intra-patient molecular-clinical therapy correlations are impossible.

Without the critical mass of tissue and data necessary to identify optimal molecular targets for lung cancer and drugs active against these targets, new discoveries that offer the only hope of long-term survival for many lung cancer patients remain elusive.

This study facilitates the collection of biospecimens from advanced lung cancer patients and routine determination of a panel of documented clinically significant biomarkers. In addition, it will centrally integrate and standardize research tissue samples with corresponding proteomic, genomic, molecular and clinical data across a multitude of institutions and oncology networks

ELIGIBILITY:
Inclusion Criteria:

* M1A or B NSCLC with any number of prior therapies or any stage Small cell Lung Cancer (SCLC) with any number of prior therapies
* Planned systemic therapy (i.e. intent to treat)
* Provision of written informed consent for biospecimen storage, broad genetic and proteomic analysis of tumor and normal tissues, without restrictions, AND correlation with outcome data
* Aged 18 years and over.
* Measurable or evaluable disease.
* ECOG performance status of 0-2 with expected survival of at least 3 months.
* Tumor specimens:
* Tumor specimens:
* 4.7.1 First Priority: availability of a minimum of a 1 X 10 mm core fresh frozen tumor, or ≥3 mm diameter spherical pellet from a pleural effusion (≥50% tumor cells), or ≥3 mm diameter spherical pellet from a fine needle aspirate (≥50% tumor cells) from clinically indicated interventional procedures, with no systemic anti-cancer therapy or radiation to all sites of evaluable disease between collection of the biopsy and entry into the study (e.g. if a brain metastasis was radiated but the lung tumor was not, then the latter could still be biopsied and the subject enrolled after radiation therapy of the brain metastasis (and vice versa)).

or

* Second Priority: availability of paraffin-embedded tumor (via biopsies or pleural effusions) at least 5 X 5 mm (3 X 3 mm for pleural effusions) cross-sectional tumor area, with no systemic anti-cancer therapy or radiation to all sites of evaluable disease between collection of the biopsy and entry into the study; the collection of the paraffin-embedded tissues may have taken place up to 12 months prior to enrollment in CASTLE.
* Willingness to undergo all study collection procedures and sample analyses including prerequisite baseline molecular testing via ResponseDX: Lung (Response Genetics Inc.) and VeriStrat (Biodesix) - see 6.3 below for details.
* Exclusion criteria
* Other co-existing malignancies except for basal cell carcinoma or cervical cancer in situ.
* Compromise of patient diagnosis or staging if tissue is harvested for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced stage lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2010-11; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Collect, process, store, and distribute for peer-reviewed research studies tumor-related and normal biospecimens from advanced stage lung cancer patients | 7 years

SECONDARY OUTCOMES:
Maintain a centralized, computerized database of all specimens | 7 years
  Database would contain uniform and complete demographic, pathologic, and clinical information
Facilitate integration of molecular assays and other laboratory studies with clinical patient outcomes | 7 years
Enable the discovery of novel genes and proteins related to cancer and its therapies | 7 years
  Obtain funding from National Institutes of Health based on use of the biorepository

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Addario Lung Cancer Medical Institute - CASTLE — http://alcmi.net/research/castle-study/